CLINICAL TRIAL: NCT06695221
Title: Improving Health Outcomes With Kefir
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00139307
Record Dates: First submitted 2024-11-13; First posted 2024-11-19 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Systemic Inflammatory Response; Diabetes Mellitus, Type 2; Cardiovascular Diseases
Keywords: Kefir; Systemic inflammation; Vascular markers; Gut microbiota; Fermented Foods
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Milk

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants living with T2D (Experimental): Randomly assigned to consume either traditional kefir or milk as a placebo.
  Interventions: Dietary Supplement: Traditional Kefir; Dietary Supplement: Milk (placebo)
- Participants with higher risk of T2D (Experimental): Randomly assigned to consume either traditional kefir or milk as a placebo.
  Interventions: Dietary Supplement: Traditional Kefir; Dietary Supplement: Milk (placebo)

INTERVENTIONS:
Dietary Supplement: Traditional Kefir — 350 mL/day of traditional fermented/prepared kefir
Dietary Supplement: Milk (placebo) — 350 mL/day of commercial 2% fat milk

SUMMARY:
The purpose of the study is to ascertain whether traditional kefir not only enhances vascular health but also contributes to improved immune outcomes in both male and female participants at higher risk or living with Type 2 Diabetes (T2D) after 12 weeks of treatment.

DETAILED DESCRIPTION:
Participants who sign the written consent form will undergo a screening process to determine eligibility for study entry. At the baseline visit, recruited participants will be randomized in a double-blind manner (participant and study coordinator) to consume either 350 mL of traditional fermented kefir or 350 mL of a placebo (milk) daily. During the 12 weeks of intervention, health outcomes will be measured and collected for further analysis.

ELIGIBILITY:
Inclusion Criteria:

1. females and males (24-70 years old) living in Edmonton (or Edmonton area/driving distance);
2. overweight or obesity (BMI >25 Caucasian, >23 Asian);
3. at higher risk of T2D (fasting blood glucose ≥ 5.6 - 6.9 mmol/L or/and HbA1C ≥ 5.5 - 6.4%); or
4. with diagnosis of T2D (fasting blood glucose ≥ 7.0 mmol/L or/and HbA1C ≥ 6.5%).

Exclusion Criteria:

1. a usual high intake (maximum intake 3 servings/week) of fermented foods excluding cheese (i.e., kefir, kombucha, kimchi, etc.) for the past 3 months;
2. gastrointestinal (GI) disorders of any kind;
3. being pregnant or breastfeeding;
4. monogenic dyslipidemias and endocrine disorders except for diabetes;
5. use of medications within the last 3 months (i.e., antibiotics or antifungals, corticosteroids, methotrexate, or immunosuppressive cytotoxic agents);
6. any health conditions deemed to interfere with primary outcomes at the investigator's discretion (e.g., kidney disease, liver disease, cancer, GI surgery, heavy alcohol consumption, etc.);
7. having a pacemaker or any electrical medical device that prevents the individual from undergoing the bioelectrical impedance analysis bioimmunoassay (BIA) test."

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Glycated Hemoglobin (HbA1c) Levels (Percentage) | Baseline, 6 weeks, 12 weeks
  The primary outcome is the change in HbA1c levels, measured as a percentage of total hemoglobin using standard laboratory methods. This measurement assesses average blood glucose levels over the past 2-3 months, providing insight into the effect of our traditional kefir on long-term glucose regulation.

SECONDARY OUTCOMES:
Change in Fasting Plasma Glucose Levels (mmol/L) | Baseline, 6 weeks, 12 weeks
  This outcome measures the change in fasting plasma glucose levels using standard blood glucose analysis. The assessment at multiple time points will provide insights into the short-term impact of our traditional kefir on fasting glucose regulation.
Change in Total Cholesterol (mmol/L) | Baseline, 6 weeks, 12 weeks
  This outcome evaluates changes in total cholesterol concentration, providing insights into the effect of our traditional kefir on lipid metabolism and cardiovascular risk. It will be measured in serum samples using standard laboratory methods.
Change in Low-Density Lipoprotein Cholesterol (LDL-C) (mmol/L) | Baseline, 6 weeks, 12 weeks
  This outcome measures the change in LDL-C levels, a primary marker of cardiovascular health, to assess the potential cardiovascular benefits of our traditional kefir. It will be measured in serum samples using standard laboratory methods.
Change in High-Density Lipoprotein Cholesterol (LDL-C) (mmol/L) | Baseline, 6 weeks, 12 weeks
  This outcome assesses the change in HDL-C concentration to evaluate whether our traditional kefir consumption has beneficial effects on lipid profiles. It will be measured in serum samples using standard laboratory methods.
Change in Triglyceride levels (mmol/L) | Baseline, 6 weeks, 12 weeks
  This outcome measures the change in triglyceride concentration to determine the effect of our traditional kefir on lipid metabolism and metabolic health. It will be measured in serum samples using standard laboratory methods.
Change in Circulating C-Reactive Protein (CRP) Levels (mg/L) | Baseline, 6 weeks, 12 weeks
  This outcome measures changes in CRP, a systemic inflammation marker, providing insight into whether our traditional kefir impacts inflammatory responses in participants. It will be measured in plasma samples using standard laboratory methods.
Change in Interleukin-2 (IL-2) in Supernatant of Ex Vivo Stimulated Cells from Whole Blood (pg/mL) | Baseline, 6 weeks, 12 weeks
  This outcome measures changes in IL-2 levels in the supernatant of ex vivo-stimulated cells derived from whole blood, serving as a surrogate marker of T-cell proliferation. IL-2 will be quantified using cytokine analysis of cell culture supernatants following mitogen stimulation. This assessment provides insight into immune function and response.
Change in T Helper Cell Response Measured by Interferon-Gamma (IFN-γ) Levels in Supernatant of Ex Vivo Stimulated Cells from Whole Blood (pg/mL) | Baseline, 6 weeks, 12 weeks
  This outcome evaluates changes in interferon-gamma (IFN-γ) levels in the supernatant of ex vivo-stimulated cells derived from whole blood. IFN-γ is a key cytokine secreted by T helper cells, serving as an indicator of cellular immune response and Th1 activity. IFN-γ will be quantified using cytokine analysis of cell culture supernatants following mitogen stimulation.
Change in Tumor Necrosis Factor-Alpha (TNF-α) Levels in Supernatant of Ex Vivo Stimulated Cells from Whole Blood (pg/mL) | Baseline, 6 weeks, 12 weeks
  This outcome measures changes in TNF-α levels in the supernatant of ex vivo-stimulated cells derived from whole blood. TNF-α is a pro-inflammatory cytokine and serves as a marker of immune system activation. TNF-α will be quantified using cytokine analysis of cell culture supernatants following mitogen stimulation.
Change in Gut Microbiome Composition and Functional Capacity (Relative Abundance) | Baseline, 6 weeks, 12 weeks
  This outcome examines changes in the composition and functional capacity of the gut microbiome using 16S rRNA gene sequencing or metagenomic analysis. The analysis will focus on relative abundance and diversity of bacterial taxa and functional pathways associated with metabolic health.

OTHER OUTCOMES:
Changes in Body Weight (Kg) | Baseline, 6 weeks, 12 weeks
  This outcome measures changes in body weight using a calibrated digital scale. Participants' weight will be assessed while wearing light clothing and no shoes. This measurement evaluates the effect of our traditional kefir on overall body mass.
Change in Body Mass Index (BMI) (kg/m²) | Baseline, 6 weeks, 12 weeks
  BMI will be calculated using body weight (kg) and height (m) measurements. Height will be measured using a stadiometer at baseline only, and BMI will be monitored to assess changes in body composition.
Change in Waist Circumference (cm) | Baseline, 6 weeks, 12 weeks
  This outcome evaluates changes in waist circumference, measured at the umbilical level using a non-elastic tape. This measurement serves as an indicator of central adiposity and fat distribution.
Change in Hip Circumference (cm) | Baseline, 6 weeks, 12 weeks
  Hip circumference will be measured at the widest part of the hips using a non-elastic tape. This outcome helps determine changes in fat distribution and body shape.
Change in Body Composition (Percentage of Fat Mass and Fat-Free Mass) Measured by Bioelectrical Impedance Analysis (BIA) | Baseline, 6 weeks, 12 weeks
  Body composition will be assessed using BIA to determine changes in fat mass and fat-free mass as percentages of total body weight. Participants will be measured in a fasted state with consistent hydration levels for accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Wastyk HC, Fragiadakis GK, Perelman D, Dahan D, Merrill BD, Yu FB, Topf M, Gonzalez CG, Van Treuren W, Han S, Robinson JL, Elias JE, Sonnenburg ED, Gardner CD, Sonnenburg JL. Gut-microbiota-targeted diets modulate human immune status. Cell. 2021 Aug 5;184(16):4137-4153.e14. doi: 10.1016/j.cell.2021.06.019. Epub 2021 Jul 12. PMID 34256014
- [Background] Savaiano DA, Hutkins RW. Yogurt, cultured fermented milk, and health: a systematic review. Nutr Rev. 2021 Apr 7;79(5):599-614. doi: 10.1093/nutrit/nuaa013. PMID 32447398
- [Background] Braga Tibaes JR, Barreto Silva MI, Makarowski A, Cervantes PB, Richard C. The nutrition and immunity (nutrIMM) study: protocol for a non-randomized, four-arm parallel-group, controlled feeding trial investigating immune function in obesity and type 2 diabetes. Front Nutr. 2023 Sep 1;10:1243359. doi: 10.3389/fnut.2023.1243359. eCollection 2023. PMID 37727636
- [Background] Bourrie BC, Willing BP, Cotter PD. The Microbiota and Health Promoting Characteristics of the Fermented Beverage Kefir. Front Microbiol. 2016 May 4;7:647. doi: 10.3389/fmicb.2016.00647. eCollection 2016. PMID 27199969
- [Background] Bourrie, B, Cotter, P, Willing, BP, 2018. Traditional kefir reduces weight gain and improves plasma and liver lipid profiles more successfully than a commercial equivalent in a mouse model of obesity. Journal of Functional Foods, 46: 29-37. https://doi.org/10.1016/j.jff.2018.04.039
- [Background] Bourrie BCT, Richard C, Willing BP. Kefir in the Prevention and Treatment of Obesity and Metabolic Disorders. Curr Nutr Rep. 2020 Sep;9(3):184-192. doi: 10.1007/s13668-020-00315-3. PMID 32472367
- [Background] Bourrie BCT, Ju T, Fouhse JM, Forgie AJ, Sergi C, Cotter PD, Willing BP. Kefir microbial composition is a deciding factor in the physiological impact of kefir in a mouse model of obesity. Br J Nutr. 2021 Jan 28;125(2):129-138. doi: 10.1017/S0007114520002743. Epub 2020 Jul 20. PMID 32684173
- [Background] Bourrie BCT, Forgie AJ, Ju T, Richard C, Cotter PD, Willing BP. Consumption of the cell-free or heat-treated fractions of a pitched kefir confers some but not all positive impacts of the corresponding whole kefir. Front Microbiol. 2022 Nov 24;13:1056526. doi: 10.3389/fmicb.2022.1056526. eCollection 2022. PMID 36504827
- [Background] Bourrie BCT, Forgie AJ, Makarowski A, Cotter PD, Richard C, Willing BP. Consumption of kefir made with traditional microorganisms resulted in greater improvements in LDL cholesterol and plasma markers of inflammation in males when compared to a commercial kefir: a randomized pilot study. Appl Physiol Nutr Metab. 2023 Sep 1;48(9):668-677. doi: 10.1139/apnm-2022-0463. Epub 2023 May 24. PMID 37224566